CLINICAL TRIAL: NCT06409611
Title: MUSCLE EFFECTS OF NEUROMUSCULAR ELECTROSTIMULATION IN MECHANICALLY VENTILATED PATIENTS IN AN ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Jose Roberto Lapa e Silva, Full Professor of Pneumology, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07071995
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Unit Acquired Weakness
Keywords: neuromuscular electrical stimulation; Intensive Care Unit Acquired Weakness

STUDY DESIGN:
Intervention Model Description: fes/parametros
Who Masked: Outcomes Assessor
Masking Description: olhar em artigos
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neuromuscular electrical stimulation (NMES) (Experimental): For the NMES group, NMES therapy will be performed for 1 hour, once a day and for 10 days. Using the following parameters: Biphasic and symmetrical rectangular pulse, with a frequency of 50Hz, pulse width of 500μs, ON time of 10 seconds, OFF time of 15 seconds, 3 seconds of rise time and 2 seconds of descent time. The intensity is increased to the point that there is complete muscle contraction, visible or palpable. The maximum intensity will be 120 mA.
  Interventions: Device: neuromuscular electrical stimulation
- Placebo (Active Comparator): This group will perform conventional physiotherapy according to institutional protocol. Rehabilitation was oriented towards achieving daily motor milestones (sitting on the edge of the bed, sitting in an armchair, getting up and walking) according to the CPAx scale. The same electrostimulation device will be installed, but it will not be turned on.
  Interventions: Device: neuromuscular electrical stimulation

INTERVENTIONS:
Device: neuromuscular electrical stimulation — Application of neuromuscular electrical stimulation using the NeuroDyn III device (IBRAMED, Amparo - SP)

SUMMARY:
To prevent the development of ICUAW, both early mobilization and neuromuscular electrical stimulation (NMES) have been shown to prevent muscle atrophy in critically ill patients by preserving muscle mass. Furthermore, it is of great value that muscle assessment using kinesiological ultrasound becomes routine to monitor this patient's profile with regard to strength, muscle quality and muscle mass. Our objective is to evaluate the muscular changes promoted by NMES in patients under mechanical ventilation. This is a randomized clinical trial study, which will perform NMES sessions for at least 10 days in mechanically ventilated patients. They will also undergo ultrasound assessments of the quadriceps. Patients will be divided into a control group and an NMES group. In addition, general information recorded in the medical record will be collected, such as basic characteristics, laboratory tests and general assessments.

DETAILED DESCRIPTION:
This is a randomized clinical trial study, which will be carried out at the Hospital Universitário Pedro Ernesto between the months of May 2024 and November 2025, where patients admitted to the General CTI will undergo muscle assessments through ultrasound and a protocol of NMES over a period of 10 days. Participants will be randomized and allocated into 2 groups: placebo and NMES. After randomization, general information recorded in the medical record will be collected, such as baseline characteristics, laboratory tests, general assessments, Sequential Organ Failure Assessment Score (SOFA), Chelsea Critical Care Physical Assessment Tool (CPAx) functional scale, edema classification, quality and type of contraction during each NMES session, days on pressure support ventilation (PSV) and pressure or volume assist-controlled ventilation (PCV or VCV), use of neuromuscular blocker, corticosteroids, vasoactive amine and the type and days of diet. Patients will undergo ultrasound evaluation of the pennation angle (AP) of the vastus lateralis, cross-sectional area (CSA) of the rectus femoris, thickness (ESP) of the quadriceps and echogenicity (ECHO) of the rectus femoris, within the first 24h post intubation, at 5 days and 10 days post intubation. Muscle assessment was carried out by professional physiotherapists trained and certified for this purpose. For the NMES group, NMES therapy will be performed for 1 hour, once a day and for 10 days. Using the following parameters: Biphasic and symmetrical rectangular pulse, with a frequency of 50Hz, pulse width of 500μs, ON time of 10 seconds, OFF time of 15 seconds, 3 seconds of rise time and 2 seconds of descent time. The intensity is increased to the point that there is complete muscle contraction, visible or palpable. The maximum intensity will be 120 mA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. On mechanical ventilation in the first 24 hours;
3. Provision of written, informed and/or agreed consent for a family member.

Exclusion Criteria:

1. Trauma to the lower limb;
2. History of neurological, neuromuscular or debilitating diseases;
3. Spinal cord injury;
4. Rhabdomyolysis;
5. Vascular insufficiency or amputation of the lower limb;
6. Previous immobility;
7. Epilepsy;
8. Musculoskeletal and skin conditions or situations that may interfere in conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pennation angle (degrees) | First, fifth and tenth days.
  Pennation angle measured by ultrasound

SECONDARY OUTCOMES:
Cross-sectional area (cm2) | First, fifth and tenth days.
  Cross-sectional area (cm2) measured by ultrasound
Echogenicity (AU) | First, fifth and tenth days.
  Echogenicity (AU) measured by ultrasound
Thickness (cm) | First, fifth and tenth days.
  Thickness (cm) measured by ultrasound
Days free from mechanical ventilation | 28-day interval.
  Days free from mechanical ventilation within a 28-day interval.
Extubation success rate (%) | 28-day interval.
  Extubation success rate (%)
ICU mortality rate (%). | 28-day interval.
  ICU mortality rate (%).

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Pedro Ernesto University Hospital, Rio de Janeiro, Rio de Janeiro
  - State University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Universidade do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No